CLINICAL TRIAL: NCT00347165
Title: Intravitreal Bevacizumab Therapy for Neovascular Age-Related Macular Degeneration: A Pilot Study
Brief Title: Intravitreal Bevacizumab for Age-Related Macular Degeneration
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: undefined
Sponsor: Asociación para Evitar la Ceguera en México (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AvastinDMRE
Record Dates: First submitted 2006-06-29; First posted 2006-07-04 (Estimated); Last update posted 2024-05-30 (Actual); Status verified 2024-05

CONDITIONS: Age Related Macular Degeneration
Keywords: macular degeneration; angiogenesis; antibodies
MeSH Terms: conditions — Macular Degeneration | interventions — Bevacizumab

INTERVENTIONS:
Drug: bevacizumab intravitreal injection

SUMMARY:
The purpose of this study is to determine whether intravitreal injection of bevacizumab is effective in the treatment of neovascular age related macular degeneration

DETAILED DESCRIPTION:
The neovascular age related macular degeneration(AMD) is a important cause of legal blindness in adults older than 50 years. Currently the treatment is photodynamic therapy that offer stabilization and limited visual improvement after 2 years of therapy. Bevacizumab has been reported effective used as intravenous injection for AMD. But serious side effects have been reported with the use of this drug in oncologic patients. The intravitreal use has been reported in limited case reports and safety and efficacy should be determined.

The purpose of this study is efficacy and safety of 2.5 mg intravitreal of bevacizumab for AMD

ELIGIBILITY:
Inclusion Criteria:

* age >50 age related macular degeneration

Exclusion Criteria:

* moderate to severe cataract glaucoma intraocular surgery diabetes mellitus non controlled hypertension coronary artery disease

Ages: 50 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2005-09 (Actual); Primary Completion 2006-06 (Actual); Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
Improvement of visual acuity at 6 months

SECONDARY OUTCOMES:
Retinal thickness at 6 months
Leakiness in fluorangiography at 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Hugo Quiroz-Mercado, MD, Study Chair — Asociación para Evitar la Ceguera en México
Locations (1):
- Hospital Luis Sanchez Bulnes, Mexico City, Mexico City, Mexico

REFERENCES:
- [Background] Rosenfeld PJ, Moshfeghi AA, Puliafito CA. Optical coherence tomography findings after an intravitreal injection of bevacizumab (avastin) for neovascular age-related macular degeneration. Ophthalmic Surg Lasers Imaging. 2005 Jul-Aug;36(4):331-5. PMID 16156152